CLINICAL TRIAL: NCT01384487
Title: Comparative Study of the Nidek Optical Coherence Tomography RS-3000 and the RTVue OCT Predicate Device for the Measurements of Retinal and RNFL Thickness, Optic Disc Analysis, Pachymetry, Anterior Chamber Imaging and SLO Imaging.
Brief Title: Nidek RS3000 Comparative Study
Status: Completed | Type: Observational
Sponsor: Nidek Co. LTD. (Industry)
Responsible Party: Sponsor
Other Study IDs: Nidek RS3000-1
Record Dates: First submitted 2011-06-27; First posted 2011-06-29 (Estimated); Last update posted 2012-02-20 (Estimated); Status verified 2012-02

CONDITIONS: Glaucoma; Retinal Disease; Corneal Disease
Keywords: Viewing and axial cross sectional imaging of ocular; structures, including the anterior chamber
MeSH Terms: conditions — Glaucoma; Retinal Diseases; Corneal Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Normal Eyes: Eyes without disease
- Eyes with Glaucoma
- Eyes with Retinal Disease
- Eyes with Corneal Disease: Including post keratorefractive surgery

SUMMARY:
The primary objective of this clinical study is to compare the Nidek RS-3000 Optical Coherence Tomography (OCT) device to the Optovue RTVue OCT. The secondary objective is to evaluate any adverse events found during the clinical study.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects of legal age and who have full legal capacity to volunteer on the date the informed consent is signed.
2. Subjects who follow the instructions by Principal/Clinical Investigator or clinical staff at the clinical site, and can visit on a scheduled examination date.
3. Subjects who sign an informed consent form to participate in the clinical study.
4. Subjects who agree to take the qualifying examination and RS-3000 and RTVue data acquisition.

Exclusion Criteria:

1. Diabetes mellitus (DM) and/or diabetic retinopathy
2. Hypertension (HT)
3. Cerebral infarction, cerebral hemorrhage, cranial nerve neoplasm and other central nervous system diseases affecting vision
4. Cardiac, hepatic, renal and hematologic diseases
5. Current systemic administration of steroid
6. History of anticancer agent etc.
7. Optically-stimulated epileptic seizure
8. Dementia
9. Subjects who have other life threatening and debilitating systemic diseases

NOTE: Additional detailed inclusion/exclusion ophthalmic criteria dependent upon study population also exist

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2011-06; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Total Retinal Thickness | One Visit
Inner Retinal Thickness | One Visit
Outer Retinal Thickness | One Visit
RNFL Thickness | One Visit
Optic Disc Analysis | One Visit
G Chart | One Visit
Anterior Chamber Angle Image | One Visit
SLO Image | One Visit
Pachymetry | One Visit

SECONDARY OUTCOMES:
Any adverse events | One Visit

CONTACTS AND LOCATIONS:
Overall Officials: Robert Weinreb, M.D., Principal Investigator — UCSD, Hamilton Glaucoma Center
Locations (1):
- Hamilton Glaucoma Center, La Jolla, California, United States